CLINICAL TRIAL: NCT00540228
Title: Immunogenicity, Safety and Reactogenicity of GSK Biologicals' Influenza Vaccine GSK1247446A With Various Formulations in Subjects Aged 18-64 Years
Brief Title: Study to Evaluate an Influenza Vaccine Candidate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 110794; 2007-003776-18 (EudraCT Number)
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Results first posted 2013-04-30 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Influenza
Keywords: Influenza; Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant

ARMS (5):
- GSK1247446A 1 Group (Experimental): Subjects aged 18-64 years at the time of enrolment received 1 dose of GSK1247446A with a full dose of AS03 adjuvant at Day 0. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Influenza Vaccine GSK1247446A - 4 different formulations
- GSK1247446A 2 Group (Experimental): Subjects aged 18-64 years at the time of enrolment received 1 dose of GSK1247446A with 1/2 dose of AS03 adjuvant at Day 0. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Influenza Vaccine GSK1247446A - 4 different formulations
- GSK1247446A 3 Group (Experimental): Subjects aged 18-64 years at the time of enrolment received 1 dose of GSK1247446A with 1/4 dose of AS03 adjuvant at Day 0. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Influenza Vaccine GSK1247446A - 4 different formulations
- GSK1247446A 4 Group (Experimental): Subjects aged 18-64 years at the time of enrolment received 1 dose of GSK1247446A with 1/8 dose of AS03 adjuvant at Day 0. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Influenza Vaccine GSK1247446A - 4 different formulations
- Fluarix Group (Active Comparator): Subjects aged 18-64 years at the time of enrolment received 1 dose of FluarixTM at Day 0. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: Influenza Vaccine GSK1247446A - 4 different formulations — Single dose, Intramuscular injection
  Arms: GSK1247446A 1 Group; GSK1247446A 2 Group; GSK1247446A 3 Group; GSK1247446A 4 Group
Biological: Fluarix™ — Single dose, Intramuscular injection
  Arms: Fluarix Group

SUMMARY:
In order to find the formulation leading to a maximal increase of the immune response while maintaining an acceptable safety profile, this study is designed to evaluate the immunogenicity, safety and reactogenicity of the different formulations of GSK Biologicals' influenza vaccine administered in adults aged 18-64 years.

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects who the investigator believes that they can and will comply with the requirements of the protocol .
* A male or female between, and including, 18 - 64 years of age at the time of vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must have a negative pregnancy test, practice adequate contraception for 30 days prior to vaccination, and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within three months prior to the first vaccine dose
* Administration of a vaccine not foreseen by the study protocol from 30 days before vaccination, up to 21 days after vaccination.
* History of hypersensitivity to a previous dose of influenza vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s)
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Confirmed influenza infection within a year preceding the study start.
* Administration of an influenza vaccine within a year preceding the study start.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Concurrent participation in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Acute disease at the time of enrolment.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.
* History of administration of experimental/licensed vaccine containing squalene and/or tocopherol within the last 12 months.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1006 (Actual)
Dates: Start 2007-10-05 (Actual); Primary Completion 2008-05-08 (Actual); Study Completion 2008-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- France (5):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Lagord
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Germany (5):
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 110794 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110794 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110794 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110794 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110794 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110794 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Started | 200 | 198 | 204 | 202 | 202
Completed | 197 | 197 | 204 | 202 | 202
Not Completed | 3 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group | Total
Number analyzed (Participants) | 200 | 198 | 204 | 202 | 202 | 1006
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.5 (14.14) | 40.3 (13.79) | 39.7 (14.37) | 39.7 (14.31) | 40.1 (14.11) | 40.1 (14.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 116 | 115 | 140 | 123 | 609
  Male | 85 | 82 | 89 | 62 | 79 | 397

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The 3 influenza strains assessed were A/Solomon Islands (SOLO), A/Wisconsin (WISC) and B/Malaysia (MALA). The seropositivity cut-off assay was 1:10. The results for Day 0 and Day 21 are the primary efficacy variables.
Time Frame: At Days 0, 21 and 180
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning Immunogenicity outcomes variables were available and for whom assay results were available for antibodies against at least one study vaccine component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 189 | 190 | 192 | 192 | 187
titers
  SOLO, Day 0 [N=187;189;190;192;185] | 13.0 [10.9 to 15.5] | 12.3 [10.2 to 14.8] | 12.9 [10.6 to 15.8] | 14.9 [12.3 to 18.2] | 15.1 [12.5 to 18.2]
  SOLO, Day 21 [N=187;189;190;192;185] | 203.2 [171.7 to 240.3] | 155.8 [128.2 to 189.4] | 164.9 [137.6 to 197.8] | 151.1 [124.7 to 183.1] | 191.0 [158.5 to 230.2]
  SOLO, Day 180 [N=189;190;192;192;187] | 81.3 [68.3 to 96.8] | 71.1 [58.8 to 86.1] | 76.3 [63.2 to 92.0] | 80.7 [66.7 to 97.5] | 97.6 [82.5 to 115.5]
  WISC, Day 0 [N=187;189;190;192;185] | 29.4 [23.8 to 36.4] | 30.0 [24.3 to 37.2] | 29.9 [24.5 to 36.5] | 27.2 [22.6 to 32.8] | 37.4 [30.2 to 46.4]
  WISC, Day 21 [N=187;189;190;192;185] | 380.1 [321.3 to 449.8] | 326.4 [275.6 to 386.7] | 319.9 [270.0 to 379.1] | 273.9 [232.0 to 323.3] | 335.3 [286.2 to 392.7]
  WISC, Day 180 [N=189;190;192;192;187] | 174.3 [145.6 to 208.8] | 149.5 [125.3 to 178.3] | 164.0 [138.0 to 195.0] | 133.0 [112.5 to 157.3] | 176.2 [151.7 to 204.6]
  MALA, Day 0 [N=187;189;190;192;185] | 25.8 [21.3 to 31.3] | 27.3 [22.6 to 32.9] | 22.6 [18.8 to 27.1] | 23.2 [19.5 to 27.8] | 27.0 [22.2 to 32.7]
  MALA, Day 21 [N=187;189;190;192;185] | 225.8 [195.3 to 261.1] | 246.1 [210.9 to 287.2] | 195.5 [165.1 to 231.4] | 171.2 [144.2 to 203.2] | 217.8 [184.3 to 257.4]
  MALA, Day 180 [N=189;190;192;192;187] | 106.6 [91.7 to 124.0] | 119.6 [103.7 to 138.0] | 97.2 [83.2 to 113.5] | 95.7 [82.1 to 111.7] | 108.8 [93.1 to 127.0]

2. Secondary Outcome: Number of Seroconverted Subjects Against 3 Strains of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a four-fold increase in post-vaccination titer. The 3 influenza strains assessed were A/Solomon Islands (SOLO), A/Wisconsin (WISC) and B/Malaysia (MALA).
Time Frame: At Days 21 and 180
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 189 | 190 | 192 | 192 | 187
subjects
  SOLO, Day 21 [N=187;189;190;192;185] | 154 | 141 | 133 | 119 | 131
  SOLO, Day 180 [N=189;190;192;192;187] | 117 | 108 | 102 | 102 | 110
  WISC, Day 21 [N=187;189;190;192;185] | 150 | 147 | 142 | 142 | 118
  WISC, Day 180 [N=189;190;192;192;187] | 112 | 97 | 112 | 106 | 100
  MALA, Day 21 [N=187;189;190;192;185] | 136 | 127 | 128 | 127 | 125
  MALA, Day 180 [N=189;190;192;192;187] | 99 | 99 | 98 | 102 | 88

3. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against 3 Strains of Influenza Disease.
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0. The 3 influenza strains assessed were A/Solomon Islands (SOLO), A/Wisconsin (WISC) and B/Malaysia (MALA).
Time Frame: At Days 21 and 180
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 189 | 190 | 192 | 192 | 187
fold increase
  SOLO, Day 21 [N=187;189;190;192;185] | 15.6 [12.7 to 19.2] | 12.7 [10.2 to 15.8] | 12.8 [10.1 to 16.1] | 10.1 [8.0 to 12.8] | 12.7 [9.9 to 16.2]
  SOLO, Day 180 [N=189;190;192;192;187] | 6.4 [5.3 to 7.7] | 5.9 [4.8 to 7.2] | 5.9 [4.8 to 7.2] | 5.4 [4.4 to 6.7] | 6.5 [5.2 to 8.0]
  WISC, Day 21 [N=187;189;190;192;185] | 12.9 [10.5 to 16.0] | 10.9 [8.9 to 13.3] | 10.7 [8.6 to 13.2] | 10.1 [10.1 to 12.3] | 9.0 [7.2 to 11.2]
  WISC, Day 180 [N=189;190;192;192;187] | 6.0 [5.0 to 7.2] | 5.0 [4.2 to 6.1] | 5.4 [4.5 to 6.6] | 4.9 [4.1 to 5.9] | 4.7 [3.9 to 5.8]
  MALA, Day 21 [N=187;189;190;192;185] | 8.7 [7.2 to 10.6] | 9.0 [7.3 to 11.2] | 8.7 [7.0 to 10.8] | 7.4 [6.1 to 8.9] | 8.1 [6.6 to 9.9]
  MALA, Day 180 [N=189;190;192;192;187] | 4.2 [3.5 to 4.9] | 4.4 [3.6 to 5.3] | 4.4 [3.6 to 5.3] | 4.1 [3.5 to 4.8] | 4.0 [3.3 to 4.8]

4. Secondary Outcome: Number of Seroprotected Subjects Against 3 Strains of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:40. The 3 influenza strains assessed were A/Solomon Islands (SOLO), A/Wisconsin (WISC) and B/Malaysia (MALA).
Time Frame: At Days 0, 21 and 180
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 189 | 190 | 192 | 192 | 187
subjects
  SOLO, Day 0 [N=187;189;190;192;185] | 45 | 46 | 43 | 52 | 50
  SOLO, Day 21 [N=187;189;190;192;185] | 177 | 170 | 169 | 166 | 172
  SOLO, Day 180 [N=189;190;192;192;187] | 157 | 144 | 144 | 151 | 159
  WISC, Day 0 [N=187;189;190;192;185] | 90 | 90 | 96 | 91 | 95
  WISC, Day 21 [N=187;189;190;192;185] | 183 | 186 | 185 | 184 | 183
  WISC, Day 180 [N=189;190;192;192;187] | 175 | 175 | 175 | 173 | 183
  MALA, Day 0 [N=187;189;190;192;185] | 80 | 88 | 81 | 86 | 88
  MALA, Day 21 [N=187;189;190;192;185] | 183 | 186 | 180 | 180 | 178
  MALA, Day 180 [N=189;190;192;192;187] | 174 | 177 | 167 | 171 | 169

5. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against 4 Strains of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs). The 4 influenza strains assessed were A/Wisconsin (WISC), B/Malaysia (MALA), A/Brisbane (BRIS) and B/Florida (FLOR). The seropositivity cut-off assay was 1:28.
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 47 | 48 | 44 | 47 | 42
titers
  WISC, Day 0 [N=43;47;44;43;42] | 134.3 [94.6 to 190.8] | 136.3 [101.4 to 183.1] | 160.8 [111.0 to 232.9] | 148.0 [107.0 to 204.5] | 212.5 [138.2 to 326.6]
  WISC, Day 21 [N=47;48;44;47;42] | 1193.7 [876.6 to 1625.5] | 859.6 [637.8 to 1158.5] | 1027.9 [760.3 to 1389.8] | 842.3 [641.9 to 1105.2] | 864.0 [654.2 to 1140.9]
  MALA, Day 0 [N=46;48;44;44;42] | 34.1 [25.7 to 45.1] | 36.5 [25.9 to 51.3] | 33.3 [24.4 to 45.4] | 27.7 [21.1 to 36.2] | 49.7 [35.2 to 70.0]
  MALA, Day 21 [N=44;48;43;42;42] | 162.5 [117.6 to 224.5] | 161.5 [128.6 to 202.9] | 141.0 [103.8 to 191.3] | 130.5 [98.7 to 172.7] | 166.0 [111.2 to 247.7]
  BRIS, Day 0 [N=47;48;44;47;41] | 494.2 [389.0 to 627.7] | 365.9 [298.3 to 449.0] | 392.5 [319.1 to 482.8] | 445.7 [369.2 to 538.0] | 466.8 [355.2 to 613.5]
  BRIS, Day 21 [N=47;48;44;47;42] | 1151.5 [901.8 to 1470.4] | 847.5 [668.0 to 1075.3] | 884.2 [673.2 to 1161.2] | 1038.2 [799.3 to 1348.6] | 867.1 [658.9 to 1141.1]
  FLOR, Day 0 [N=45;48;44;47;42] | 48.9 [35.2 to 67.9] | 56.9 [38.6 to 83.9] | 51.0 [35.2 to 73.9] | 46.8 [32.7 to 66.9] | 76.7 [51.1 to 115.3]
  FLOR, Day 21 [N=43;48;43;43;42] | 94.3 [68.8 to 129.3] | 113.6 [79.7 to 162.0] | 92.1 [60.6 to 139.9] | 82.7 [57.9 to 118.2] | 131.1 [93.3 to 184.2]

6. Secondary Outcome: Geometric Mean of Influenza-specific Cluster of Differentiation (CD) 4 T-cells.
Description: The mean was calculated for CD4 T-cells (per million CD4 T-cells) producing at least two different cytokines (All Doubles), at least CD40L, at least INF gamma (IFN-γ), at least IL2 and at least TNF alpha (TNF-α).
Time Frame: At Days 0, 21 and 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 46 | 47 | 43 | 47 | 41
cells
  All Doubles, Day 0 [N=45;47;43;47;39] | 2106.16 (1274.90) | 2043.17 (894.18) | 2252.44 (1726.88) | 2103.66 (1370.89) | 1976.23 (1051.16)
  All Doubles, Day 21 [N=45;45;40;45;39] | 3857.76 (2195.47) | 3366.93 (1693.40) | 3103.30 (1549.21) | 2827.84 (1561.60) | 2489.15 (1468.71)
  All Doubles, Day 180 [N=46;42;42;43;41] | 2628.96 (1353.46) | 2249.88 (1325.73) | 1963.38 (1245.21) | 2153.12 (1473.45) | 1952.02 (1240.63)
  CD40L, Day 0 [N=45;47;43;47;39] | 1914.96 (1241.38) | 1863.96 (830.55) | 2045.86 (1638.11) | 1954.13 (1290.77) | 1827.67 (1033.38)
  CD40L, Day 21 [N=45;45;40;45;39] | 3337.89 (1982.59) | 2947.20 (1487.13) | 2624.30 (1316.60) | 2472.98 (1378.17) | 2223.74 (1398.63)
  CD40L, Day 180 [N=46;42;42;43;41] | 2108.04 (1190.42) | 1758.95 (1093.80) | 1581.31 (1184.99) | 1731.00 (1331.05) | 1560.76 (1009.77)
  IFN-γ, Day 0 [N=45;47;43;47;39] | 1379.33 (987.07) | 1377.13 (741.31) | 1510.84 (1349.58) | 1342.57 (1040.63) | 1260.97 (809.24)
  IFN-γ, Day 21 [N=45;45;40;45;39] | 2525.91 (1615.78) | 2233.24 (1371.05) | 2056.40 (1205.90) | 1824.69 (1265.29) | 1565.79 (1064.31)
  IFN-γ, Day 180 [N=46;42;42;43;41] | 1792.74 (1075.76) | 1546.55 (1055.94) | 1335.62 (970.49) | 1440.09 (1199.84) | 1299.95 (894.25)
  IL2, Day 0 [N=45;47;43;47;39] | 1684.24 (983.48) | 1657.28 (744.17) | 1796.33 (1354.89) | 1732.91 (1140.54) | 1572.69 (812.49)
  IL2, Day 21 [N=45;45;40;45;39] | 3020.09 (1741.78) | 2634.64 (1415.24) | 2343.15 (1199.20) | 2256.02 (1251.58) | 1933.10 (1153.35)
  IL2, Day 180 [N=46;42;42;43;41] | 2121.67 (1088.48) | 1816.26 (1116.55) | 1571.19 (987.96) | 1797.79 (1228.49) | 1581.73 (1028.49)
  TNF-α, Day 0 [N=45;47;43;47;39] | 1606.64 (1087.17) | 1522.70 (747.67) | 1712.42 (1355.23) | 1548.00 (1094.03) | 1421.82 (781.48)
  TNF-α, Day 21 [N=45;45;40;45;39] | 2767.02 (1598.41) | 2337.38 (1068.82) | 2109.45 (1075.51) | 1990.60 (1157.58) | 1639.31 (975.93)
  TNF-α, Day 180 [N=46;42;42;43;41] | 1980.39 (1078.92) | 1654.90 (944.90) | 1454.40 (898.01) | 1627.67 (1155.63) | 1392.05 (933.32)

7. Secondary Outcome: Geometric Mean of Influenza-specific Cluster of Differentiation (CD) 8 T-cells.
Description: The mean was calculated for CD8 T-cells (per million CD8 T-cells) producing at least two different cytokines (All Doubles), at least CD40L, at least INF gamma (IFN-γ), at least IL2 and at least TNF alpha (TNF-α).
Time Frame: At Days 0, 21 and 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 44 | 46 | 43 | 45 | 41
cells
  All Doubles, Day 0 [N=44;46;43;45;39] | 50.02 (113.85) | 109.63 (405.09) | 17.33 (33.12) | 64.47 (181.32) | 48.38 (82.57)
  All Doubles, Day 21 [N=44;43;40;42;38] | 47.18 (106.55) | 50.09 (101.55) | 38.53 (67.21) | 109.86 (282.04) | 55.11 (126.17)
  All Doubles, Day 180 [N=44;40;42;41;41] | 44.32 (99.11) | 126.13 (323.68) | 36.31 (95.06) | 97.27 (258.53) | 30.98 (62.35)
  CD40L, Day 0 [N=44;46;43;45;39] | 3.64 (12.37) | 5.91 (15.92) | 2.63 (8.06) | 16.27 (56.56) | 7.05 (20.43)
  CD40L, Day 21 [N=44;43;40;42;38] | 8.82 (28.38) | 10.09 (21.58) | 6.45 (16.03) | 50.83 (193.00) | 37.55 (117.41)
  CD40L, Day 180 [N=44;40;42;41;41] | 9.45 (35.59) | 15.88 (61.59) | 2.86 (8.48) | 1.68 (4.37) | 2.27 (5.83)
  IFN-γ, Day 0 [N=44;46;43;45;39] | 29.50 (53.27) | 96.91 (375.61) | 14.42 (32.92) | 44.80 (137.59) | 17.31 (38.50)
  IFN-γ, Day 21 [N=44;43;40;42;38] | 24.86 (61.18) | 48.07 (106.65) | 25.65 (49.98) | 64.98 (178.63) | 32.11 (104.54)
  IFN-γ, Day 180 [N=44;40;42;41;41] | 38.18 (50.84) | 110.75 (303.91) | 20.62 (47.56) | 79.85 (239.36) | 19.80 (37.25)
  IL2, Day 0 [N=44;46;43;45;39] | 35.59 (91.49) | 75.41 (309.22) | 8.81 (16.65) | 46.22 (130.46) | 43.59 (81.53)
  IL2, Day 21 [N=44;46;43;45;39] | 36.98 (85.05) | 21.51 (42.47) | 31.28 (59.89) | 87.86 (244.84) | 50.84 (116.74)
  IL2, Day 180 [N=44;40;42;41;41] | 27.36 (87.59) | 74.03 (183.59) | 24.50 (82.62) | 57.15 (136.73) | 28.73 (55.08)
  TNF-α, Day 0 [N=44;46;43;45;39] | 42.98 (109.79) | 102.72 (391.96) | 15.42 (28.60) | 54.73 (156.41) | 46.18 (91.78)
  TNF-α, Day 21 [N=44;43;40;42;38] | 37.93 (109.46) | 44.16 (99.17) | 31.55 (59.52) | 90.48 (239.47) | 37.82 (110.79)
  TNF-α, Day 180 [N=44;40;42;41;41] | 34.70 (86.94) | 111.10 (299.67) | 33.60 (80.50) | 79.54 (208.13) | 25.63 (56.06)

8. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms.
Description: Assessed solicited local symptoms were ecchymosis, pain, redness and swelling at injection site. Any = incidence of a particular symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal everyday activity. Grade 3 redness/swelling/ecchymosis = redness/swelling/ecchymosis spreading beyond 50 millimeters (mm) of the injection site.
Time Frame: During the 7-day (Days 0-6) post vaccination period
Population: The analysis was based on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 200 | 198 | 204 | 202 | 202
subjects
  Any Ecchymosis | 11 | 9 | 8 | 14 | 7
  Grade 3 Ecchymosis | 1 | 0 | 0 | 1 | 1
  Any Pain | 182 | 175 | 167 | 151 | 121
  Grade 3 Pain | 5 | 5 | 3 | 1 | 1
  Any Redness | 75 | 66 | 53 | 64 | 49
  Grade 3 Redness | 17 | 4 | 3 | 2 | 2
  Any Swelling | 69 | 54 | 49 | 48 | 27
  Grade 3 Swelling | 11 | 4 | 5 | 3 | 2

9. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [oral temperature above (>) 38.0 degrees Celsius (°C)], headache, myalgia, nausea and shivering. Any = incidence of a particular symptom regardless of grade intensity or relationship with the study vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0°C. Related = symptom considered by the investigator to have a causal relationship to study vaccination.
Time Frame: During the 7-day (Days 0-6) post vaccination period
Population: The analysis was based on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 200 | 198 | 204 | 202 | 202
subjects
  Any Arthralgia | 64 | 51 | 38 | 39 | 25
  Grade 3 Arthralgia | 4 | 4 | 2 | 0 | 1
  Related Arthralgia | 52 | 49 | 32 | 31 | 20
  Any Fatigue | 103 | 90 | 86 | 78 | 47
  Grade 3 Fatigue | 5 | 4 | 2 | 2 | 2
  Related Fatigue | 81 | 83 | 72 | 62 | 34
  Fever >38°C | 27 | 16 | 8 | 6 | 3
  Fever ≥ 39°C | 2 | 0 | 0 | 0 | 0
  Related Fever | 23 | 13 | 8 | 6 | 3
  Any Headache | 90 | 77 | 68 | 66 | 51
  Grade 3 Headache | 7 | 2 | 4 | 3 | 1
  Related Headache | 72 | 61 | 49 | 49 | 36
  Any Myalgia | 102 | 85 | 74 | 70 | 49
  Grade 3 Myalgia | 6 | 6 | 4 | 0 | 2
  Related Myalgia | 81 | 77 | 59 | 57 | 40
  Any Nausea | 25 | 28 | 12 | 13 | 11
  Grade 3 Nausea | 1 | 2 | 3 | 0 | 0
  Related Nausea | 19 | 22 | 10 | 11 | 6
  Any Shivering | 74 | 53 | 40 | 34 | 12
  Grade 3 Shivering | 4 | 5 | 1 | 1 | 2
  Related Shivering | 64 | 50 | 31 | 29 | 8

10. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Medically Significant Conditions (MSCs).
Description: MSCs were defined as conditions prompting emergency room visits or physician visits that were not related to common diseases or routine visits. Any = incidence of a particular symptom regardless of grade intensity or relationship with the study vaccination. Grade 3 = event which prevented normal activities. Related = event assessed by the investigator as causally related to the study vaccination
Time Frame: From Day 0 to Day 180
Population: The analysis was based on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 200 | 198 | 204 | 202 | 202
subjects
  Subjects with any MSCs | 70 | 56 | 53 | 64 | 45
  Subjects with grade 3 and related MSCs | 2 | 2 | 0 | 0 | 1
  Subjects with related MSCs | 5 | 2 | 0 | 0 | 1

11. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = any unsolicited AE regardless of intensity or relationship to vaccination. Grade 3 = unsolicited AE that prevented normal activity Related = unsolicited AE assessed by the investigator as related to the vaccination.
Time Frame: During the 21-day (Days 0-20) post vaccination period
Population: The analysis was based on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 200 | 198 | 204 | 202 | 202
subjects
  Subjects with any AE(s) | 85 | 91 | 70 | 82 | 80
  Subjects with grade 3 AE(s) | 4 | 10 | 3 | 10 | 5
  Subjects with related AE(s) | 37 | 41 | 25 | 19 | 14

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 to Day 180
Population: The analysis was based on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
Number analyzed (Participants) | 200 | 198 | 204 | 202 | 202
subjects | 7 | 3 | 3 | 4 | 2

ADVERSE EVENTS:
Time Frame: SAE(s)reports were collected during the entire study period (Day 0 - Day 180); Solicited local and general symptoms: during the 7-day (Days 0-6) follow-up period after any vaccination, Unsolicited AE(s): during the 21-day follow-up period (Days 0 to 20) after any vaccination.
Description: For this study, the Total Number (#) of Participants Affected by Other (non-serious) Adverse Events (AEs) was analyzed separately for expected AEs and for unexpected AEs. A consolidated analysis of all expected and unexpected AEs was not technically possible to be performed and the relevant data are no longer available. Therefore, the Total #Participants Affected in Other Adverse Events Table is currently populated by the highest value of #Participants affected within other AE's table.
Arm/Group | GSK1247446A 1 Group | GSK1247446A 2 Group | GSK1247446A 3 Group | GSK1247446A 4 Group | Fluarix Group
All-Cause Mortality (participants affected / at risk) | 1/200 | 0/198 | 0/204 | 0/202 | 0/202
Serious Adverse Events (participants affected / at risk) | 7/200 | 3/198 | 3/204 | 4/202 | 2/202
Other Adverse Events (participants affected / at risk) | 182/200 | 175/198 | 167/204 | 151/202 | 121/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1247446A 1 Group (N=200) | GSK1247446A 2 Group (N=198) | GSK1247446A 3 Group (N=204) | GSK1247446A 4 Group (N=202) | Fluarix Group (N=202)
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1247446A 1 Group (N=200) | GSK1247446A 2 Group (N=198) | GSK1247446A 3 Group (N=204) | GSK1247446A 4 Group (N=202) | Fluarix Group (N=202)
Ecchymosis (General disorders) | 11 | 9 | 8 | 14 | 7
Pain (General disorders) | 182 | 175 | 167 | 151 | 121
Redness (General disorders) | 75 | 66 | 53 | 64 | 49
Swelling (General disorders) | 69 | 54 | 49 | 48 | 27
Arthralgia (General disorders) | 64 | 51 | 38 | 39 | 25
Fatigue (General disorders) | 103 | 90 | 86 | 78 | 47
Fever >38°C (General disorders) | 27 | 16 | 8 | 6 | 3
Headache (General disorders) | 90 | 77 | 68 | 66 | 51
Myalgia (General disorders) | 102 | 85 | 74 | 70 | 49
Nausea (General disorders) | 25 | 28 | 12 | 13 | 11
Shivering (General disorders) | 74 | 53 | 40 | 34 | 12
Headache (Nervous system disorders) | 14 | 12 | 16 | 19 | 14
Rhinitis (Infections and infestations) | 5 | 8 | 6 | 9 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.